CLINICAL TRIAL: NCT05833399
Title: Assessment of the Inter-patient Variability in Clinical Response and Correlated Genetic Variations in Substance Use Disorders
Brief Title: Correlation of Genetic Variations With Clinical Response in Substance Use Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: INTERPAT-VAR-ClinResp-SUD-1
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Substance Use Disorders; Substance Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Quetiapine Fumarate; Olanzapine; Mirtazapine; Carbamazepine; Sertraline; Amitriptyline; Chlorpromazine; Risperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Addicted patients on treatment with psychiatric medications.: Addicted patients receiving treatment with either quetiapine, olanzapine, mirtazapine, carbamazepine, sertraline, amitriptyline, chlorpromazine or risperidone as oral dosage forms of usual prescribed doses for psychiatric disorders.
  Interventions: Drug: Quetiapine, olanzapine, mirtazapine, carbamazepine, sertraline, amitriptyline, chlorpromazine and risperidone
- Healthy non-addicted controls.: Individuals who have never been addicted to any substance of use and did not receive any treatment with psychiatric medications.

INTERVENTIONS:
Drug: Quetiapine, olanzapine, mirtazapine, carbamazepine, sertraline, amitriptyline, chlorpromazine and risperidone — Medications are prescribed orally for outpatient or inpatient treatment of addicted patients.
  Other Names: Seroquel, Olapex, Remeron, Tegretol, Moodapex, Tryptizol, Neurazine and Apexidone.
  Groups: Addicted patients on treatment with psychiatric medications.

SUMMARY:
This research outcomes can be summarized as follows:

1. Pharmacogenomic analysis of Substance Use Disorder (SUD) and medications used for the treatment of SUD.
2. Identification of novel genetic variations related to SUD specifically in the Egyptian population.
3. Validation of currently known genetic variations associated with SUD. When the functional interpretation of common or rare variants in studied genes becomes available, such pharmacogenomic information can be used to improve pharmacotherapy individualization.

DETAILED DESCRIPTION:
This is a correlational cross-sectional study to investigate the correlation of some genetic variants to the predisposition to SUD in addicted patients as well as to the clinical response of the medications they receive as a part of their treatment plan.

Subjects participating in this study are those receiving outpatient or inpatient programs for the management of SUD with or without psychiatric disorders, supported by the specialized mental health care facility; "Al-Maa'moura Hospital for Psychiatry" in Alexandria.

An informed consent is obtained from each participant prior their contribution to the study. Approval from the General Secretariat of Mental Health and Addiction Treatment (GSMHAT), Ministry of Health and Population (MoHP), has been obtained before conducting the study as well as from the Ethics Committee, Faculty of Medicine, Alexandria University.

A minimal total sample size of 100 participants with SUD, male or female, and another 40 controls will be included in the study. This sample size was calculated with the assistance of instructors in the Department of Medical Statistics, Medical Research Institute, Alexandria University. The targeted sample is selected regarding the inclusion and exclusion criteria.

Patients' medical records will be checked to select the medications of interest. The medications selected include those most prescribed by the psychiatrists assigned at the hospital. They include quetiapine, carbamazepine, amitriptyline, olanzapine, sertraline, chlorpromazine, risperidone, and mirtazapine.

A structured questionnaire will be designed for proper patient data collection. It will be validated for its content using the jury method. The reliability, internal consistency of the questionnaire, will be estimated through the calculated value of Cronbach's alpha. Face to face interviewing with the eligibly selected patients will be done after they sign the patient consent. The questionnaire will be divided into sectors regarding the patients' sociodemographic data, their general health condition, their SUD, and the medications they receive for treatment.

Blood samples will be collected from controls and patients receiving their treatment. These samples will be used for preparation of plasma in which the drug levels will be estimated. They will also be used for isolation of DNA to screen selected mutations, sequence selected genes or perform whole genome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Addicted patients receiving outpatient or inpatient treatment for SUD with or without psychiatric disorders at a mental health care facility.

Exclusion Criteria:

* Patients with renal or hepatic impairment.
* Patients receiving chemotherapy or radiotherapy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects participating in this study are those receiving outpatient or inpatient programs for the management of SUD with or without psychiatric disorders, supported by the specialized mental health care facility; "Al-Maa'moura Hospital for Psychiatry" in Alexandria, Egypt.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacogenomic analysis of SUD and medications used for the treatment of SUD. | 1 year

SECONDARY OUTCOMES:
Identification of novel genetic variations related to SUD specifically in the Egyptian population. | 1 year

OTHER OUTCOMES:
Validation of currently known genetic variations associated with SUD. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M El-Gowilly, PhD, Principal Investigator — Professor of Pharmacology and Toxicology, Alexandria University; Ahmed F El-Yazbi, PhD, Principal Investigator — Professor of Pharmacology and Toxicology, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Lecturer of Clinical Pharmacy and Pharmacy Practice, Alexandria University; Nefertiti A El-Nikhely, PhD, Principal Investigator — Associate Professor of Biochemistry, Alexandria University; Aymen H Hamouri, MSc, Principal Investigator — Psychiatrist Consultant
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided